CLINICAL TRIAL: NCT01601288
Title: Prospective Database of All Patients Who Have Undergone Pulmonary Function Testing at Singapore General Hospital
Brief Title: Database of All Patients Who Have Undergone Pulmonary Function Testing at Singapore General Hospital
Status: Completed | Type: Observational
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2011/845/Cpftdatabase
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Obstructive Pulmonary Diseases; Restrictive Lung Disease; Cough; Dyspnea
Keywords: obstructive lung disease; restrictive lung disease; cough; dyspnea
MeSH Terms: conditions — Lung Diseases, Obstructive; Cough; Dyspnea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to create a prospective database of all patients who have undergone pulmonary function testing from which the investigators can study the clinical phenotypes of various respiratory conditions. The investigators hope by understanding the differences in these myriad phenotypes to be able to provide individualized, patient-targeted therapy in the future.

DETAILED DESCRIPTION:
Recent studies have shown that clinical phenotyping of patients with various respiratory conditions is important in the understanding of the disease process, clinical response to treatment, and prognosis. Pulmonary function testing is a very important aspect of clinical phenotyping in many respiratory conditions. Creating a database will enable us to study the various phenotypes within each respiratory condition. This will allow us to better understand each disease, with a view to provide personalized patient care targeted at their specific phenotype and hence better clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1) All patients who have undergone pulmonary function testing at the Singapore General Hospital pulmonary function laboratory

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Prospective data collection of all patients who have undergone pulmonary function testing at Singapore General Hospital
Sampling Method: Non-Probability Sample
Enrollment: 17000 (Actual)
Dates: Start 2012-05; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Diagnoses based on pulmonary function test interpretation | 7 days
  Interpretation of pulmonary function tests by a certified respiratory physician

CONTACTS AND LOCATIONS:
Overall Officials: Su Ying Low, BMBCh, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Background] Nishimura M, Makita H, Nagai K, Konno S, Nasuhara Y, Hasegawa M, Shimizu K, Betsuyaku T, Ito YM, Fuke S, Igarashi T, Akiyama Y, Ogura S; Hokkaido COPD Cohort Study Investigators. Annual change in pulmonary function and clinical phenotype in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2012 Jan 1;185(1):44-52. doi: 10.1164/rccm.201106-0992OC. PMID 22016444
- [Background] Nathan SD, Shlobin OA, Weir N, Ahmad S, Kaldjob JM, Battle E, Sheridan MJ, du Bois RM. Long-term course and prognosis of idiopathic pulmonary fibrosis in the new millennium. Chest. 2011 Jul;140(1):221-229. doi: 10.1378/chest.10-2572. PMID 21729893